CLINICAL TRIAL: NCT04968158
Title: Confirmatory Efficacy and Safety Study of the Fixed-dose Combination of Etoricoxib / Tramadol Versus Acetaminophen / Tramadol for the Management of Acute Low Back Pain.
Brief Title: Efficacy and Safety of Fixed-dose Combination of Etoricoxib/Tramadol vs Acetaminophen/Tramadol for Acute Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIL-30138-III-21(1)
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Acute Low Back Pain
Keywords: Back pain; Etoricoxib; Tramadol; Fixed dose
MeSH Terms: conditions — Back Pain | interventions — Etoricoxib; Tramadol; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Etoricoxib/Tramadol (Experimental): Administered orally, one packet of etoricoxib / tramadol granules diluted in 100 ml of water, every 24 hours for 7 days.
  Interventions: Drug: Etoricoxib 90 mg / Tramadol 50 mg
- Group B: Acetaminophen / Tramadol (Active Comparator): Administered orally, one tablet, every 8 hours, for 7 days.
  Interventions: Drug: Acetaminophen 325 mg / Tramadol 37.5 mg

INTERVENTIONS:
Drug: Etoricoxib 90 mg / Tramadol 50 mg — One packet diluted in 100 ml of water, every 24 hours of 90 mg/50 mg.
  Other Names: E/T
  Arms: Group A: Etoricoxib/Tramadol
Drug: Acetaminophen 325 mg / Tramadol 37.5 mg — One tablet, every 8 hours of 325 mg/ 37.5 m
  Other Names: A/T
  Arms: Group B: Acetaminophen / Tramadol

SUMMARY:
Phase IIIb, longitudinal, multicenter, randomized, open-label clinical trial to evaluate the efficacy and safety of the fixed-dose combination of etoricoxib 90 mg and tramadol 50 mg compared with fixed-dose therapy of acetaminophen 325 mg and tramadol 37.5 mg for the management of acute low back pain.

DETAILED DESCRIPTION:
Patients with back pain from the level of the lowest rib to the gluteal crease, with or without radiation to the legs, as a first-time episode or after another at least 6 months before and lasting no more than 6 weeks, that in the opinion of the doctor requires treatment with the combination of an anti-inflammatory and an analgesic. Study to evaluate the efficacy and safety of the fixed-dose combination of etoricoxib 90 mg and tramadol 50 mg compared with the fixed-dose therapy of acetaminophen 325 mg and tramadol 37.5 mg for the management of acute low back pain. Evaluate and compare the average change in pain reported through the VAS at 3, 5 and 7 days with respect to its baseline measurement by treatment group. An exploratory analysis of the data will be carried out to identify aberrant, outliers, or missing values. To present the numerical variables, the measures of central tendency and dispersion appropriate to the distribution of the data will be used and the categorical variables will be expressed as frequency and percentage.

ELIGIBILITY:
Inclusion Criteria:

* Any sex.
* That the subject agree to participate in the study and give informed consent in writing.
* Age> 18 years and ≤ 60 years of age at the beginning of the study.
* Diagnosis of acute low back pain as a first-time episode or after another episode, maximum 6 months before and lasting no more than 6 weeks.
* Patient with low back pain reported as moderate to severe intensity (VAS> 4 cm).
* Women of childbearing age who have an acceptable contraceptive method (eg barrier, oral hormonal, injectable, subdermal).

Exclusion Criteria:

* Patients in whom the study drug is contraindicated for medical reasons.
* Patients with an allergy or hypersensitivity to the active principle, study drugs, related products or excipients.
* Positive pregnancy test, women who are pregnant, breastfeeding or planning a pregnancy while conducting the study.
* A significant history of gastrointestinal disorders (for example: Gastric ulcer, Crohn's disease, Ulcerative Colitis, etc.).
* Previous treatment with opioids and / or NSAIDs (Non-Steroidal Anti-Inflammatory Drugs) reported in the medical history in the last 72 hours at study entry.
* Patients with a history of alcohol or drug abuse in the last year according to DSM-V (Diagnostic and Statistical Manual of Mental Disorders).
* Patients who are receiving monoamine oxidase inhibitors (MAOIs) or who have received them within the past 2 weeks.
* Patients with a history of established ischemic heart disease, peripheral arterial disease and / or cerebrovascular disease (including patients who have recently undergone coronary artery bypass grafting or angioplasty).
* Patients with status epileptic seizure disorders and grand mal seizures.
* Patients with a history of severe acute or chronic liver failure.
* Patients with a history of moderate to severe renal failure.
* Patient with a history of chronic pain (eg, fibromyalgia, Paget's disease, bone pain induced by metastatic cancer).
* Low back pain due to major trauma (eg vertebral fracture, post-traumatic spondylolisthesis), or due to a visceral disorder (eg dysmenorrhea, endometriosis).
* At medical criteria, a disease that affects the prognosis and prevents outpatient management, for example, but not restricted to: intestinal obstruction, paralytic ileus, end-stage cancer, kidney, heart, respiratory or liver failure or mental illness or with surgical procedures or scheduled hospitals.
* History / presence of any disease or condition that, in the Investigator's opinion, could pose a risk to the patient or confuse the efficacy and safety of the study results. ----Patients with symptoms suggesting an active COVID-19 infection (i.e., fever, cough, dyspnea) and / or contact in the past 14 days with a suspected or positive COVID-19 patient.
* Oncological patients (except basal cell skin cancer) or with serious diseases that, in the opinion of the investigator, have a serious prognosis or a life expectancy of less than 1 year, as well as mental illnesses.
* The patient is participating in another clinical study involving an investigational treatment or participated in one in the previous 4 weeks.
* Patients whose participation in the study may be influenced (employment relationship with the research center or sponsor, inmates, etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Average change in reported pain | Baseline, 3, 5 and 7 days.
  Compare the average change in pain reported through the VAS (Visual Analog Scale) per treatment group. In a straight 10 centimeter line in which one end means no pain and the other end means the worst pain imaginable, the participants mark the amount of pain feeling at that moment

SECONDARY OUTCOMES:
Proportion of patients with a 30% reduction in pain intensity | Baseline and 7 days.
  Describe the proportion of patients who reported a 30% reduction in pain intensity measure by the VAS (Visual Analog Scale) per treatment group. In a straight 10 centimeter line in which one end means no pain and the other end means the worst pain imaginable, the participants mark the amount of pain feeling at that moment.
Degree of disability due to low back pain | Baseline and 7 days.
  Evaluate the degree of disability due to low back pain measured through the Oswestry disability scale per treatment group. It measures the limitations in daily activities in the presence of pain in the lumbar region, consists of 10 questions with 6 possible answers considering the intensity of the pain, basic activities of daily life such as: personal care, sexual activity, sleep, travel and social life.
Degree of inability to perform daily activities | Baseline and 7 days.
  Assess the degree of inability to perform daily activities through the Roland-Morris scale per group. It´s a self-applied scale where the extreme values range between 0 (absence of disability) and 24 (maximum disability) and is categorized according to the relevance of the score obtained where the optimal threshold of variation is 3 and 4 points.
Adverse events | 7 days.
  Compare the frequency of adverse events presented during the study between the treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Zurqui Ramírez, M.D, Principal Investigator — Icaro Investigación en Medicina S.A. de C.V.; Adelfia Urenda Quezada, M.D, Principal Investigator — Mediadvance Clinical S.A.P.I. de Quezada; Alejandro González Rebatu y González, M.D, Principal Investigator — Clinical Research Institute S.C.
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Soto-Padilla M, Espinosa-Mendoza RL, Sandoval-Garcia JP, Gomez-Garcia F. [Comparative study between plate-graft, cage-plate and peek cage in cervical arthrodesis for cervical stenosis]. Acta Ortop Mex. 2015 Jan-Feb;29(1):40-5. Spanish. PMID 26999925
- [Background] Casser HR, Seddigh S, Rauschmann M. Acute Lumbar Back Pain. Dtsch Arztebl Int. 2016 Apr 1;113(13):223-34. doi: 10.3238/arztebl.2016.0223. PMID 27120496
- [Background] Guevara-Lopez U, Covarrubias-Gomez A, Elias-Dib J, Reyes-Sanchez A, Rodriguez-Reyna TS; Consensus Group of Practice Parameters to Manage Low Back Pain. Practice guidelines for the management of low back pain. Consensus Group of Practice Parameters to Manage Low Back Pain. Cir Cir. 2011 May-Jun;79(3):264-79, 286-302. English, Spanish. PMID 22381000
- [Background] Gonzalez Maza C, Moscoso Lopez L, Ramirez Elizalde G, Abdo Andrade A. [Multimodal treatment of chronic unspecific low back pain]. Acta Ortop Mex. 2010 Mar-Apr;24(2):88-94. Spanish. PMID 20831016
- [Background] Chandanwale AS, Sundar S, Latchoumibady K, Biswas S, Gabhane M, Naik M, Patel K. Efficacy and safety profile of combination of tramadol-diclofenac versus tramadol-paracetamol in patients with acute musculoskeletal conditions, postoperative pain, and acute flare of osteoarthritis and rheumatoid arthritis: a Phase III, 5-day open-label study. J Pain Res. 2014 Aug 12;7:455-63. doi: 10.2147/JPR.S67817. eCollection 2014. PMID 25152629
- [Background] Bravo L, Mico JA, Berrocoso E. Discovery and development of tramadol for the treatment of pain. Expert Opin Drug Discov. 2017 Dec;12(12):1281-1291. doi: 10.1080/17460441.2017.1377697. Epub 2017 Sep 17. PMID 28920461
- [Background] Dhillon S. Tramadol/paracetamol fixed-dose combination: a review of its use in the management of moderate to severe pain. Clin Drug Investig. 2010;30(10):711-38. doi: 10.2165/11205830-000000000-00000. PMID 20701403
- [Background] Subedi M, Bajaj S, Kumar MS, Yc M. An overview of tramadol and its usage in pain management and future perspective. Biomed Pharmacother. 2019 Mar;111:443-451. doi: 10.1016/j.biopha.2018.12.085. Epub 2018 Dec 27. PMID 30594783
- [Derived] Zuqui-Ramirez MA, Belalcazar-Lopez VM, Urenda-Quezada A, Gonzalez-Rebatu Y Gonzalez A, Sander-Padilla JG, Lugo-Sanchez LA, Rodriguez-Vazquez IC, Rios-Brito KF, Arguedas-Nunez MM, Canales-Vazquez E, Gonzalez-Canudas J. Multimodal Analgesia Approach in Acute Low Back Pain Management: A Phase III Study of a Novel Analgesic Combination of Etoricoxib/Tramadol. Pain Ther. 2024 Dec;13(6):1511-1528. doi: 10.1007/s40122-024-00653-y. Epub 2024 Sep 10. PMID 39256291
- See also: World Health Organization. Musculoskeletal disorders [Internet]. Descriptive notes. 2019. — http://www.who.int/es/news-room/fact-sheets/detail/musculoskeletal-conditions
- See also: "That establishes the tests and procedures to demonstrate that a drug is interchangeable. Requirements to which the Authorized Third Parties that carry out the interchangeability tests must be ". — http://www.dof.gob.mx/nota_detalle.php?codigo=5314833&fecha=20/09/2013
- See also: "Installation and operation of pharmacovigilance: This document establishes the guidelines on which pharmacovigilance activities must be carried out" — http://dof.gob.mx/nota_detalle.php?codigo=5490830&fecha=19/07/2017
- See also: "That establishes the criteria for the execution of research projects for health in human beings" — http://dof.gob.mx/nota_detalle.php?codigo=5284148&fecha=04/01/2013